CLINICAL TRIAL: NCT03660579
Title: Beer or Ethanol Effects on the Response to High Intensity Interval Training: A Controlled Study in Healthy Individuals: BEER - HIIT Study
Brief Title: Beer or Ethanol Effects on the Response to High Intensity Interval Training: A Controlled Study in Healthy Individuals
Acronym: BEER-HIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Manuel Castillo Garzón, University Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 321/CEIH/2017
Record Dates: First submitted 2018-07-20; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Drinking, Alcohol; Exercise
Keywords: Physical fitness; Recovery; Stress; Training; HIIT; Beer
MeSH Terms: conditions — Alcohol Drinking; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- HIIT-CON (No Intervention): No intervention: Control
- HIIT-AB Group (Experimental): Intake:
  330ml (women) or 2x300 ml (men) of beer with 5.4% alcohol. The beverage intakes will be programmed from Monday to Friday.
  Training:
  The volume in HIIT 40-65 min/week at high intensity. HIIT with short intervals. Frequency two times/week. Load variation. Gradual progression to control the exercise dose. Periodization divided in: familiarization phase, phase I, phase II. Sessions. The participants will performed 8 weight-bearing exercises (in circuit form) 2 times/set with an active rest (walking at 6 RPE scale) as many times at as defined. The HIIT intensity will controlled by RPE (0-10 RPE scale).
  All sessions will be started with a dynamic standardized warm-up, including several muscle activation exercises, and will be ended with a cooling-down protocol.
  Interventions: Other: HIIT-AB Group
- HIIT-NAB Group (Experimental): Intake:
  330 ml (women) or 2x300 ml (men) of beer without alcohol (0.0%). The beverage intakes will be programmed from Monday to Friday.
  Training:
  The volume in HIIT 40-65 min/week at high intensity. HIIT with short intervals. Frequency two times/week. Load variation. Gradual progression to control the exercise dose. Periodization divided in: familiarization phase, phase I, phase II. Sessions. The participants will performed 8 weight-bearing exercises (in circuit form) 2 times/set with an active rest (walking at 6 RPE scale) as many times at as defined. The HIIT intensity will controlled by RPE (0-10 RPE scale).
  All sessions will be started with a dynamic standardized warm-up, including several muscle activation exercises, and will be ended with a cooling-down protocol.
  Interventions: Other: HIIT-NAB Group
- HIIT-SW Group (Experimental): Intake:
  330 ml (women) or 2x300 ml (men) of sparkling water. The beverage intakes will be programmed from Monday to Friday.
  Training:
  The volume in HIIT 40-65 min/week at high intensity. HIIT with short intervals. Frequency two times/week. Load variation. Gradual progression to control the exercise dose. Periodization divided in: familiarization phase, phase I, phase II. Sessions. The participants will performed 8 weight-bearing exercises (in circuit form) 2 times/set with an active rest (walking at 6 RPE scale) as many times at as defined. The HIIT intensity will controlled by RPE (0-10 RPE scale).
  All sessions will be started with a dynamic standardized warm-up, including several muscle activation exercises, and will be ended with a cooling-down protocol.
  Interventions: Other: HIIT-SW Group
- HIIT-ASW Group (Experimental): Intake:
  330 ml (women) or 2x300 ml (men) of sparkling water with 5.4% alcohol.The beverage intakes will be programmed from Monday to Friday.
  Training:
  The volume in HIIT 40-65 min/week at high intensity. HIIT with short intervals. Frequency two times/week. Load variation. Gradual progression to control the exercise dose. Periodization divided in: familiarization phase, phase I, phase II. Sessions. The participants will performed 8 weight-bearing exercises (in circuit form) 2 times/set with an active rest (walking at 6 RPE scale) as many times at as defined. The HIIT intensity will controlled by RPE (0-10 RPE scale).
  All sessions will be started with a dynamic standardized warm-up, including several muscle activation exercises, and will be ended with a cooling-down protocol.
  Interventions: Other: HIIT-ASW Group

INTERVENTIONS:
Other: HIIT-AB Group — Group that performed HIIT and consumed 330 ml (women) or 2x300 ml (men) of beer with 5.4% alcohol.
  Arms: HIIT-AB Group
Other: HIIT-NAB Group — Group that performed HIIT and consumed 330 ml (women) or 2x300 ml (men) of beer without alcohol (0.0%).
  Arms: HIIT-NAB Group
Other: HIIT-SW Group — Group that performed HIIT and consumed the same amount of sparkling water (0.0%).
  Arms: HIIT-SW Group
Other: HIIT-ASW Group — Group that performed HIIT and consumed sparkling water with the same amount of alcohol than the pre-established beer (5.4%).
  Arms: HIIT-ASW Group

SUMMARY:
HIIT-BEER will determine the effect of habitual and moderate beer intake (330-660 ml / day, 5 days / week) on physical fitness, body composition, psychokinetic abilities and psychological status in sedentary healthy adults undergoing a HIIT training program.

DETAILED DESCRIPTION:
Aims:

To determine the effect of habitual and moderate consumption of beer on physical fitness, body composition, psychokinetic and cognitive abilities and psychological status in sedentary healthy adults undergoing a HIIT training program.

The primary hypothesis will that a HIIT program will induce an improvement on physical fitness, body composition, psychokinetic abilities and psychological responses compared to a control group but this positive effect could be blunted by alcohol intake.

Methods:

HIIT-BEER will recruit 80 sedentary, healthy, adults (50% women) aged 18-40 years.

Will be performed a 10-week controlled trial in which the effects of HIIT will be compared to a control group without training. The effects of habitual intake of different alcoholic beverage will be also compared.

After completing the baseline measurements, the selected participants will be randomly assigned to either the control or the exercise training groups. The participants included in the training groups will be asked to choose individual choice about their drinking preference for alcoholic or non-alcoholic beverages. The participants who chose alcohol intake will be randomly assigned into the training group with alcohol beer intake (5.4% Alcohol-Special Alhambra®, Cervezas Alhambra, Spain) or to the sparkling water group with exactly the same amount of distilled alcohol added. The distilled alcoholic beverage used for the investigator's study will be vodka because of the purity of its composition (37.5% ethanol and 62.5% water). The participants who chose non-alcoholic beverages will be randomized into the training groups of non-alcohol beer (0.0% alcohol-Cruzcampo®, Heineken España) or sparkling water (Eliges (IFA) Eliqua 2®, Font Salem, Spain) intakes.

So, eligible participants will be assigned to five groups: (i) a group that will performed HIIT and will consumed 330 ml (women) or 2x300 ml (men) of beer with 5.4% alcohol (HIIT-AB, n=16); (ii) a group that will performed HIIT and will consumed the same amount of beer without alcohol (0.0%) (HIIT-NAB; n=16); (iii) a group that will performed HIIT and will consumed the same amount of sparkling water (0.0%) (HIIT-W; n=16); (iv) a group that will performed HIIT and will consumed sparkling water with the same amount of alcohol than the pre-established beer (5.4%) (HIIT-ASW; n=16); and (v) a control group that will not perform any physical training program (CON; n=16).

The beverage intakes will be programmed from Monday to Friday. There will not specific recommendation for Saturday and Sunday, but the participants will be instructed to keep a moderate alcohol during the weekend.

Laboratory measures completed at baseline and 10 weeks later, include physical fitness (cardiorespiratory fitness, muscular strength), body composition, hearth rate variability (HRV), reaction time, cognitive variables and health-related questionnaires. The investigators will also obtain dietary habits data and cardiovascular disease risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40 years
* BMI:18.5-25 kg/m2
* Not engaged in regular physical activity >20min on >3days/week
* Not participating in a weight loss programme
* Stable weight over the last 5 months (body weight changes>5kg)
* Participant must be capable and willing to provide consent, understand exclusion criteria and accept the randomized group assignment
* Normal electrocardiogram
* Not personal family history related to alcohol consumption.

Exclusion Criteria:

* History of cardiovascular disease
* Diabetes
* Pregnancy or planning to get pregnant during study period
* Beta blockers or benzodiapezins use
* Taking medication for thyroid
* Other significant conditions that are life-threatening or that can interfere with or be aggravated by exercise
* Unwillingness to either complete the study requirements or to be randomized into control or training group

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Physical Fitness Cardiorespiratory fitness | Baseline and through study completion, an average of 10 weeks.
  Cardiorespiratory fitness measure through a maximum treadmill test (VO2 max.).

SECONDARY OUTCOMES:
Physical Fitness: Muscular strength (Bosco Test) | Baseline and through study completion, an average of 10 weeks.
  Muscle strength measure through: Bosco test.
Physical Fitness: Muscular strength (Handgrip strength) | Baseline and through study completion, an average of 10 weeks.
  Muscle strength measure through: Handgrip strength.
Body composition (DXA) | Baseline and through study completion, an average of 10 weeks.
  Body composition measure through: Dual-energy X-ray absorptiometry (DXA).
Body composition (Weight) | Baseline and through study completion, an average of 10 weeks.
  Body composition measure through: Anthropometry (Weight in kg).
Body composition (Height) | Baseline and through study completion, an average of 10 weeks.
  Body composition measure through: Anthropometry (Height in meter).
Body composition (Hip perimeter) | Baseline and through study completion, an average of 10 weeks.
  Body composition measure through: Anthropometry (Hip perimeter in cm)
Body composition (Waist circumference) | Baseline and through study completion, an average of 10 weeks.
  Body composition measure through: Anthropometry (Waist circumference in cm).
Body composition (Neck perimeter) | Baseline and through study completion, an average of 10 weeks.
  Body composition measure through: Anthropometry (Neck perimeter in cm).
Heart Rate Variability | Baseline and through study completion, an average of 10 weeks.
  Measure by Polar RS800CX.
Reaction time | Baseline and through study completion, an average of 10 weeks.
  Measure by Vienna Test System.
Memory | Baseline and through study completion, an average of 10 weeks.
  Measure by Spanish-Complutense Verbal Learning Test (TAVEC)
Attention | Baseline and through study completion, an average of 10 weeks.
  Measure by D2 Test.
Working Memory | Baseline and through study completion, an average of 10 weeks.
  Measure by Numbers and Letters (WISC-IV).
Verbal fluency | Baseline and through study completion, an average of 10 weeks.
  Verbal fluency assessment test.
Questionnaires and Scales | Baseline and through study completion, an average of 10 weeks.
  Measure by:
  * PREDIMED Questionnaire on Adherence to the Mediterranean Diet.
  * Beverage Intake Questionnaire (PREDIMED).
  * Questionnaire of the Five Great Factors of the Personality (BFQ).
  * Satisfaction with life (SWL).
  * Health questionnaire (SF-36).
  * International Fitness Scale Questionnaire (IFIS).
  * Beck Depression Inventory (BDI-II).
  * Life Orientation test questionnaire (LOT-R).
  * Sexual desire questionnaire.
  * Sexual functioning questionnaire.
  * Pittsburgh Sleep Quality Index.
  * Profile of Mood States Questionnaire (POMS).
  * Scale of Subjective Happiness.
  * Emotional Intelligence Scale (TMMS).
  * Scale Panas of positive and negative affect.
  * Perceived stress scale (PSS).
  * Scale of assessment of mood (EVEA).
  * Eating habits questionnaire.
  * Spanish versión of Three Factor EatingQuestionnaire-R18 (TFEQ-SP)
  * Scale of regulation of the behavior in physical exercise (BREQ-2).
  * Scale of measurement of the orientations of goals in the exercise (GOES)
Questionnaires and Scales | Every week
  Measure by:
  (BDI-II); PREDIMED Questionnaire on Adherence to the Mediterranean Diet ; Sexual desire questionnaire; Sexual functioning questionnaire; Eating habits questionnaire; Beverage Intake Questionnaire (PREDIMED); Perceived stress scale (PSS); Scale of Subjective Happiness; EVEA; IFIS; Pittsburgh Sleep Quality Index; BFQ; LOT-R; PANNAS; POMS; SWLS; TMMS-24 and TFEQ-SP.
Questionaires and Scales | Every two weeks
  Measure by:
  PSS; EVEA; PANNAS; TMMS-24
Questionnaires and Scales | Every three weeks
  Measure by:
  Scale of Subjective Happiness; Pittsburgh Sleep Quality Index; POMS; BREQ-2 and GOES.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel J. Castillo Garzón, Principal Investigator — Universidad de Granada
Locations (1):
- Universidad de Granada, Granada, Andalusia, Spain

REFERENCES:
- [Derived] Molina-Hidalgo C, De-la-O A, Dote-Montero M, Amaro-Gahete FJ, Castillo MJ. Influence of daily beer or ethanol consumption on physical fitness in response to a high-intensity interval training program. The BEER-HIIT study. J Int Soc Sports Nutr. 2020 May 27;17(1):29. doi: 10.1186/s12970-020-00356-7. PMID 32460793